CLINICAL TRIAL: NCT02111135
Title: Phase II, Observer-blind, Randomized Study on the Safety, Reactogenicity, Immunogenicity and Impact on Intestinal Shedding of a Single Dose of Monovalent High-dose Inactivated Poliovirus Type 2 Vaccine (m-IPV2 HD) or a Single Dose of Standard Trivalent Inactivated Poliovirus Vaccine (t-IPV) When Given Concomitantly With the Third Dose of Bivalent Oral Poliovirus Vaccine (b-OPV) to Infants Early in Life
Brief Title: Safety Study of a Single Dose of Monovalent High-dose Inactivated Poliovirus Type 2 Vaccine (m-IPV2 HD) in Infants Early in Life
Acronym: IPV005
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vaxtrials S.A. (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPV005ABMG
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Polio
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): b-OPV, m-IPV HD and m-OPV2
  Interventions: Biological: b-OPV; Biological: m-OPV2; Biological: m-IPV HD
- Group 2 (Active Comparator): b-OPV, t-IPV and m-OPV2
  Interventions: Biological: b-OPV; Biological: m-OPV2; Biological: t-IPV

INTERVENTIONS:
Biological: b-OPV
Biological: m-OPV2
Biological: m-IPV HD
  Arms: Group 1
Biological: t-IPV
  Arms: Group 2

SUMMARY:
Phase II, observer-blind, randomized study on the safety, reactogenicity, immunogenicity and impact on intestinal shedding of a single dose of monovalent high-dose inactivated poliovirus type 2 vaccine (m-IPV2 HD) or a single dose of standard trivalent inactivated poliovirus vaccine (t-IPV) when given concomitantly with the third dose of bivalent oral poliovirus vaccine (b-OPV) to infants early in life

ELIGIBILITY:
Inclusion Criteria:

1. Age: 6 weeks (-7 to +14 days).
2. Healthy without obvious medical conditions that preclude the subject to be in the study as established by the medical history and physical examination.
3. Written informed consent obtained from 1 or 2 parents or legal guardian as per Panama regulations.

Exclusion Criteria:

1. Previous vaccination against poliovirus.
2. Low birth weight (BW <2,500 gm).
3. Any confirmed or suspected immunosuppressive or immunodeficient condition including human immunodeficiency virus (HIV) infection.
4. Family history of congenital or hereditary immunodeficiency.
5. Major congenital defects or serious uncontrolled chronic illness (neurologic, pulmonary, gastrointestinal, hepatic, renal, or endocrine).
6. Known allergy to any component of the study vaccines.
7. Uncontrolled coagulopathy or blood disorder contraindicating intramuscular injections.
8. Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
9. Acute severe febrile illness at day of vaccination deemed by the Investigator to be a contraindication for vaccination (the child can be included at a later time if within age window and all in/exclusion criteria are met.).
10. Member of the subject's household (living in the same house or apartment unit) has received OPV in the last 3 months.
11. Subject who, in the opinion of the Investigator, is unlikely to comply with the protocol or is inappropriate to be included in the study for the safety or the benefit-risk ratio of the subject.

Ages: 6 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Safety | 6 weeks
  To assess and compare descriptively the safety of a single dose of a m-IPV2 HD vaccine in healthy infants to that of a licensed t-IPV vaccine when given concomitantly with the third dose of b-OPV measured by the incidence of serious adverse events (SAEs) and important medical events (IMEs) from the day of vaccine administration until day of last visit at study week 15 (~ week 21 of life).
Efficacy | 4 weeks
  To determine whether 1 dose of a m-IPV2 HD vaccine given to infants is superior to 1 dose of t-IPV given at study week 8 (~14 weeks of age) in inducing a humoral immune response to type 2 poliovirus when measured as seroconversion to type 2 poliovirus (type-specific titers ≥1:8 and >4-fold over expected levels of maternally-derived antibody) and as median titers four weeks later at study week 12 (~ 18 weeks of age).

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Sáez, MD, Principal Investigator — Hospital Del Niño
Locations (1):
- Hospital del Niño, Panama City, Provincia de Panamá, Panama

REFERENCES:
- [Derived] Brickley EB, Strauch CB, Wieland-Alter WF, Connor RI, Lin S, Weiner JA, Ackerman ME, Arita M, Oberste MS, Weldon WC, Saez-Llorens X, Bandyopadhyay AS, Wright PF. Intestinal Immune Responses to Type 2 Oral Polio Vaccine (OPV) Challenge in Infants Previously Immunized With Bivalent OPV and Either High-Dose or Standard Inactivated Polio Vaccine. J Infect Dis. 2018 Jan 17;217(3):371-380. doi: 10.1093/infdis/jix556. PMID 29304199
- [Derived] Saez-Llorens X, Clemens R, Leroux-Roels G, Jimeno J, Clemens SA, Weldon WC, Oberste MS, Molina N, Bandyopadhyay AS. Immunogenicity and safety of a novel monovalent high-dose inactivated poliovirus type 2 vaccine in infants: a comparative, observer-blind, randomised, controlled trial. Lancet Infect Dis. 2016 Mar;16(3):321-30. doi: 10.1016/S1473-3099(15)00488-0. Epub 2015 Dec 21. PMID 26719058